CLINICAL TRIAL: NCT04139356
Title: The Effect of Spontaneous Respiration on Pulse-oximetry Measurements and Analysis of Variability Mechanisms
Brief Title: The Effect of Spontaneous Respiration on Pulse-oximetry Measurements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Uriel Chavarria-Martinez, Professor of Internal Medicine Pulmonary and Critical Care, Universidad Autonoma de Nuevo Leon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UAutonomaNL
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Chronic Respiratory Disease; COPD; Interstitial Lung Disease
Keywords: pulseoxymetry; capnography; Dead space; cardiac output; lung recruitment; deep breaths
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: Clinical experimental trial of changes in pulse-oxymetry measurements with deep inspirations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with rest O2 desaturation (Experimental): Patient will undergo an experimental protocol consisting of 10 deep inspirations to measure and characterize changes on pulse-oxymetry values
  Interventions: Procedure: Deep breaths

INTERVENTIONS:
Procedure: Deep breaths — Patients will undergo a 6 minutes protocol. Baseline: 1 minute normal breaths. Intervention: 1 minute with 10 deep breaths, 1 each 6 secs. Pulse-oxymetry will be continuously recorded.

SUMMARY:
This is a study designed to measure, characterize and describe changes on pulse-oxymetry values produced as a result of deep breaths in patients with stable chronic hypoxemic respiratory failure.

DETAILED DESCRIPTION:
There is no standard way of measuring rest pulse-oxymetry in terms of depth of respiration. Rest pulse-oxymetry values are used in the clinical setting to make therapeutic decisions regarding the need of supplemental oxygen. The primary goal of this study is to measure the change of pulse-oxymetry values during an experimental protocol of 10 deep breaths during one minute in patients with chronic hypoxemia. 45 patients will be studied in this first phase. In a second phase, secondary goals will be to measure Vd/Vt vent, noninvasive cardiac output and CT densitometry during the same deep breaths protocol in a subset of 13 patients with the grater increase observed in the first phase of study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic lung disease causing rest hypoxemia, with rest SpO2 values equal or lower than 94% on room air
* Ambulatory patients capable of performing 6 min walking test
* Patients older than 18 years old.

Exclusion Criteria:

* Patients with significant collagen disease causing Raynaud phenomenon.
* Patients with hypothermia lower than 35 degrees Celsius
* Patients with rest SpO2 values equal or lower than 80% on room air
* Patients unable to perform PFTs
* Patients unable to complete 6 min walking test without supp O2.
* Patients unable to perform experimental deep breaths on CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in O2 saturation | Lenght of experimental protocol: 6 minutes.
  A Saturation change greater than 4% will be considered significant

SECONDARY OUTCOMES:
Vd/VT | Lenght of experimental protocol: 6 minutes.
  In a subset of 13 patients with the greater increase on O2Sat, Vd/Vt will be measured during the same protocol
Cardiac output (CO) | Lenght of experimental protocol: 6 minutes.
  In a subset of 13 patients with the greater increase on O2Sat, CO will be measured during the same protocol
CT recruitment | Lenght of experimental protocol: 6 minutes.
  In a subset of 13 patients with the greater increase on O2Sat, CT recruitment will be calculated using densitometry values during the same protocol

CONTACTS AND LOCATIONS:
Overall Officials: Uriel Chavarria, MD, Principal Investigator — Facultad de Medicina y Hospital Universitario UANL
Locations (1):
- Facultad de Medicina y Hospital Universitario UANL, Monterrey, Nuevo León, Mexico